CLINICAL TRIAL: NCT01305629
Title: Intervention Targeting Substance Using Older Adults With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: Fordham University (Other)
Responsible Party: Principal Investigator, Jeffrey T. Parsons, Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA029567-01 (NIH)
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: HIV; Medication Adherence; Substance Dependence
Keywords: HIV; Medication Adherence; Substance Use; Older adults; Treatment
MeSH Terms: conditions — Medication Adherence; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Condition (Experimental): Twelve sessions of spiritual self schema counseling, adapted to target target medication adherence and substance use.
  Interventions: Behavioral: Spiritual Self-Schema Therapy
- Education Condition (Active Comparator): Eight sessions of education with content designed to mirror the information covered in the intervention condition.
  Interventions: Behavioral: Spiritual Self-Schema Therapy

INTERVENTIONS:
Behavioral: Spiritual Self-Schema Therapy — The Spiritual Self Schema therapy (3S+) intervention will consist of a series of 12 one hour-long sessions delivered individually to participants over a four-month period. The 3S+ approach combines cognitive and behavioral therapy techniques with elements of non-theistic Buddhist philosophy to increase motivation for treatment adherence, alcohol and/or substance use reduction or abstinence and the prevention or reduction of HIV risk behaviors. 3S+ draws from self-regulation theory, self-schema theory, and self-discrepancy theory to assist participants in defining and perceiving their addict self, when their addict self is active, and its resulting negative affect state. 3S+ remediates the "addict" schema by proposing the construction of an alternate and competing schema: the "spiritual self." This spiritual self schema is compatible with HIV self-care, alcohol and drug use reduction or abstinence, adherence to treatment, and a compassionate life.

SUMMARY:
The proposed study uses a randomized controlled experimental design to evaluate the efficacy of a brief intervention using spiritual self schema (3S+) counseling to simultaneously target HIV health outcomes, and substance use among alcohol and/or drug dependent HIV positive older adults (age 50+), relative to an attention control condition. Participants will be randomly assigned to receive either: (1) 12 sessions of 3S+ counseling, adapted for the present study to target both non-injection drug use, drinking, and HIV health; or (2) 12 sessions of education about HIV health and the associated with alcohol and drug use that will serve as an attention-control.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ (provide HIV medication bottle with name on it)
* Age 50 or older (provide picture ID with DOB at baseline)
* Report current alcohol/drug dependence (AUDIT score of 8 or DAST-10 score of 4 on screener; C-DIS at baseline)
* On a prescribed HAART medication regimen and reports sub-optimal adherence (self-report missed at least 3 days in last 30 at 1 pill/day that is 90%)
* Communicate with staff and complete a survey in English or Spanish (English only for the pilot)

Exclusion Criteria:

* Current intravenous drug use (self-report at screener and baseline)
* Currently in a methadone drug treatment program (screener self-report)
* Unstable, serious psychiatric symptoms (SCID-Psych at baseline)
* Currently suicidal/homicidal (SCID-Psych at baseline)
* Gross cognitive impairment (Mini-Mental at baseline)
* Current enrollment in alcohol/drug treatment or HIV study (screener self-report)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Adherence to HIV medication | every four months over the course of a year
  Participants in the intervention condition will report greater reductions in viral load, and greater increases in CD4 counts and self-reported adherence than those in the education comparison at the end of the intervention period (4 months). Those in the intervention condition will also maintain greater reductions in viral load, and greater increases in CD4 counts and self-reported adherence than those in the education comparison condition at the three follow-up assessments (4, 8, and 12 months).
Substance use | every four months over the course of a year
  Participants in the intervention condition will report greater reductions in self-reported days of substance use and severity of dependence than those in the education comparison at at the end of the intervention period (4 months). Those in the intervention condition will also maintain greater reductions in self-reported days of substance use than those in the education comparison condition at the three follow-up assessments (4, 8, and 12 months).

SECONDARY OUTCOMES:
Mental Health/Quality of Life | every four months over the course of a year
  Participants in the intervention condition will report greater increases in mental health measures (e.g, depression, anxiety) and quality of life measures (e.g., life satisfaction, loneliness, perceived stress).
Sexual Risk | every four months over the course of a year
  Participants in the intervention condition will report greater reductions in high-risk sexual behavior compared to participants in the educational comparison condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T. Parsons, Ph.D., Principal Investigator — Hunter College, CUNY
Locations (1):
- Center for HIV/AIDS Educational Studies and Training of Hunter College, CUNY, New York, New York, United States